CLINICAL TRIAL: NCT04655066
Title: PANTHERA-Studie "Pelvic Floor Disorders in Patients Under ANtineoplastic THERApy"
Brief Title: Evaluation of the Subjectively Perceived Pelvic Floor Function in Patients With Gynecological Tumors and Breast Cancer Under Systemic Tumor Therapy Using a Validated Questionnaire
Status: Recruiting | Type: Observational
Sponsor: St. Josefs-Hospital Wiesbaden GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: PANTHERA
Record Dates: First submitted 2020-11-19; First posted 2020-12-04 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The multimodal therapy of gynecological malignancies and breast cancer often leads to an impairment of the pelvic floor function. This has a major impact on the quality of life of cancer patients. The aim of the study is to record and analyze the potential subjective impairment of the bladder, bowel and sexual function under systemic tumor therapy as well as possible influencing factors by means of validated disease-specific questionnaires. to find possible starting points for the prevention and treatment of the symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Breastcancer under tumor therapy
* Gynecological carcinoma under tumor therapy

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with gynecological tumors and breast cancer under systemic tumor therapy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 12 months
  The primary endpoint and basis for the sample size calculation is the incidence of clinically relevant deteriorations in the total score of pelvic floor function.
  Bladder function, bowel function, sedimentation problems and sexual function, QoL are recorded using scores using the validated German pelvic floor questionnaire

SECONDARY OUTCOMES:
Secondary Endpoint | 12 months
  Type of tumor (breast cancer, ovarian cancer, cervical cancer, endometrial cancer, vulvar cancer), TNM stage, body weight, height, age, type of tumor therapy, number of previous therapies (chemoline), parity, mode of delivery, nicotine abuse, medication, previous surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Josefs-Hospital Wiesbaden GmbH, Wiesbaden, Germany